CLINICAL TRIAL: NCT02951936
Title: The Utility of Regional Bioimpedance in Chronically Ventilated Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recrutment
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre Singer, Director of ICU, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A1 version 2
Record Dates: First submitted 2016-09-04; First posted 2016-11-01 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Chronic Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NiCAS treated (Experimental): Measure each patient with the NiCAS once a day If Cardiac Index < 2.9 +Total Peripheral resistance Index >3000+Mean arterial pressure >70mmHG then add vasodilators.
  If Heart Rate<60 consider to reduce beta blockers dose If Cardiac Index>4.2 and Mean arterial pressure 70-100mmHG and HR >100 then add Bata Blockers If patient have low Total Body Water then reduce diuretics If patient have High Total Body Water provide diuretics
  Interventions: Device: NiCAS treated
- Non NiCAS treated (Sham Comparator): Measure each patient with the NiCAS once a day Do note use the NiCAS parameters to direct treatment
  Interventions: Device: Non NiCAS treated

INTERVENTIONS:
Device: NiCAS treated — Measure each patient with the NiCAS once a day If Cardiac Index < 2.9 +Total Peripheral resistance Index >3000+Mean arterial pressure >70mmHG then add vasodilators.
  If Heart Rate<60 consider to reduce beta blockers dose If Cardiac Index>4.2 and Mean arterial pressure 70-100mmHG and HR >100 then add Bata Blockers If patient have low Total Body Water then reduce diuretics If patient have High Total Body Water provide diuretics
  Arms: NiCAS treated
Device: Non NiCAS treated — Measure each patient with the NiCAS once a day Do note use the NiCAS parameters to direct treatment For treatment we will use the standard care
  Arms: Non NiCAS treated

SUMMARY:
Chronically ventilated patients will be hemodynamically measured by bioimpedance (NiCAS by NI medical ltd.) for cardiac output, Total peripheral resistance and other NICAS derived parameters.

Patients fluid balance will be planned according to these parameters and the rate of liberation from ventilator and rate of worsening renal function will be measured

DETAILED DESCRIPTION:
Patients will be divided into two groups , the study group and the control group randomly assigned by a computer program .

After obtaining written informed consent , cardiac monitoring will be carried out by means of a NiCAS patients in both groups.The physician will not be exposed to the measurement data of the patients in the control group. For the research group : Monitoring will be carried out once a day , preferably at the same time the first three days . An increase in time interval is possible in accordance with an improvement in the patient . Patients will be treated according to the protocol described in Figure 1. Also , a graphic description of the various treatment zones and the exclusion zone is presented in Figure 2 .

For the control group patients will be treated according to the usual ward protocols.

The basic rules are:

Avoiding over- drying by using parameter TBW .

* Avoidance of renal dysfunction by maintaining the cardiac output above 2.3 , and avoiding the use of beta-blocker overdose in cases of low cardiac output and bradycardia as a result of maintaining an average blood pressure over 70 .
* In cases of high peripheral resistance - Reduction of resistance while maintaining normal blood pressure .

ELIGIBILITY:
Inclusion Criteria:

* All chronically ventilated patients (ventilated for more than 14 days)
* Age between 18-90

Exclusion Criteria:

* Non ventilated patient
* Total body water >80%

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
number of days ventilated | 90 days

SECONDARY OUTCOMES:
kidney function | 90 days
  will be assessed by blood test as Creatinin

IPD SHARING:
Plan to Share IPD: Yes